CLINICAL TRIAL: NCT04664569
Title: National Observatory of Bacterial Meningitis in Children and Newborns
Brief Title: National Bacterial Meningitis Study
Status: Recruiting | Type: Observational
Sponsor: Association Clinique Thérapeutique Infantile du val de Marne (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: Obs meningitis
Record Dates: First submitted 2020-12-07; First posted 2020-12-11 (Actual); Last update posted 2022-12-27 (Actual); Status verified 2022-12

CONDITIONS: Meningitis; Children, Only; Pneumococcal Conjugate Vaccine; Meningococcal Vaccines; H. Influenzae Vaccine; Neonatal Infection; Antibiotic Treatment; Case Fatality Rate
MeSH Terms: conditions — Meningitis | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort of bacterial meningitis in children
  Interventions: Other: observational study

INTERVENTIONS:
Other: observational study — observational study

SUMMARY:
Bacterial meningitis is a major cause of morbidity and mortality in childhood. Antibiotic treatment recommendations are based on epidemiological and susceptibility data. The epidemiology of bacterialméningitis has changed in recent years, mainly owing to widespread use of different conjugate vaccines. The aim of this prospective national survey is to describe epidemiology of bacteria implicated in bacterial meningitis in children.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs of meningitis, associated with positive cerebrospinal fluid (CSF) culture and/or positive CSF antigen testing (Escherichia coli K1, N. meningitidis serogroups B, A, C, Y and W-135, group B streptococci, Hib, or S. pneumoniae), and/or positive CSF polymerase chain reaction (PCR), and/or positive blood culture with CSF pleocytosis (> 10 cells/µL).
* purpura fulminans

Exclusion Criteria:

-

Ages: 0 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: children 0 day to 18 years with bacterial meningitis or purpura fulminans
Sampling Method: Non-Probability Sample
Enrollment: 8230 (Estimated)
Dates: Start 2001-01-01 (Actual); Primary Completion 2030-01-01 (Estimated); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
mortality | before the hospital discharge
  Number of death according to age and bacteria

SECONDARY OUTCOMES:
treatment failures | 48 hours after the antibiotic treatment and new lumbar puncture
  Number of antibiotic treatment failures according to bacteria after the control of lumbar puncture
impact of vaccines | before the hospital discharge
  Number of vaccination failures according to age, number of doses and bacteria

CONTACTS AND LOCATIONS:
Locations (1):
- ACTIV, Créteil, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Maunier L, Levy C, Baron A, Weill FX, Bechet S, Pardos de la Gandara M, Caseris M, Abdoul C, Dommergues MA, Cohen R, Bonacorsi S. Retrospective Description of 27 Cases of Nontyphoidal Salmonella Meningitis in Pediatrics Over 22 Years in France Pleads for a Revision of Age Limit for the Treatment of Salmonella Gastroenteritis in Children. Pediatr Infect Dis J. 2026 Jan 1;45(1):e10-e12. doi: 10.1097/INF.0000000000004966. Epub 2025 Sep 3. PMID 40924727
- [Derived] Fafi I, Cohen R, Levy C, Varon E, Amor-Chelihi L, Benhaim P, Houlier M, Koehl B, De Montalembert M, Allali S, Gauthier A, Odievre MH, Gajdos V, Escoda S, Kamdem A, Costa G, Guillaumat C, Thuret I, Ouldali N, Gaschignard J, Carbonnelle E, De Pontual L, Pham LL. High Mortality Due to Pneumococcal Meningitis in Children With Sickle Cell Disease: A French Multicenter Observational Study From 2001 to 2021. Pediatr Infect Dis J. 2025 Jun 1;44(6):496-502. doi: 10.1097/INF.0000000000004755. Epub 2025 Mar 7. PMID 40063777
- [Derived] Rybak A, Ouldali N, Varon E, Taha MK, Bonacorsi S, Bechet S, Angoulvant F, Cohen R, Levy C; French Pediatric Meningitis Network. Vaccine-preventable Pediatric Acute Bacterial Meningitis in France: A Time Series Analysis of a 19-Year Prospective National Surveillance Network. Pediatr Infect Dis J. 2024 Jan 1;43(1):74-83. doi: 10.1097/INF.0000000000004134. Epub 2023 Nov 13. PMID 38108805
- See also: Recurrent Pneumococcal Meningitis in Children: A Multicenter Case-control Study — https://pubmed.ncbi.nlm.nih.gov/31220046/
- See also: Incidence of paediatric pneumococcal meningitis and emergence of new serotypes: a time-series analysis of a 16-year French national survey — https://pubmed.ncbi.nlm.nih.gov/30049623/
- See also: Clinical and Laboratory Features of Group B Streptococcus Meningitis in Infants and Newborns: Study of 848 Cases in France, 2001-2014 — https://pubmed.ncbi.nlm.nih.gov/29045606/
- See also: Risk Factors in Children Older Than 5 Years With Pneumococcal Meningitis: Data From a National Network — https://pubmed.ncbi.nlm.nih.gov/28403047/
- See also: Neonatal Meningococcal Meningitis In France From 2001 To 2013 — https://pubmed.ncbi.nlm.nih.gov/27753774/
- See also: Comparative impact of pneumococcal conjugate vaccines on pneumococcal meningitis according to underlying conditions — https://pubmed.ncbi.nlm.nih.gov/27595445/
- See also: Outcomes of bacterial meningitis in children — https://pubmed.ncbi.nlm.nih.gov/27020729/